CLINICAL TRIAL: NCT00954161
Title: Bystander Helping Behaviour for Acute Myocardial Infarction Following a First Aid Training Programme That Draws Attention to the Barriers to Providing Help - Protocol for a Randomized Controlled Trial
Brief Title: Bystander Helping Behaviour for Myocardial Infarction Following First Aid Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Belgian Red Cross (Other); University Ghent (Other); Laerdal Medical (Industry)
Responsible Party: Bert Aertgeerts, Academic Centre for General Practice
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: S51742; S51742, ML5859, B32220096701 (Other: Commissie Medische Ethiek UZ Gasthuisberg)
Record Dates: First submitted 2009-08-06; First posted 2009-08-07 (Estimated); Last update posted 2011-05-03 (Estimated); Status verified 2011-05

CONDITIONS: Acute Myocardial Infarction
Keywords: First aid; Helping behaviour; Health education; Myocardial infarction; Emergencies
MeSH Terms: conditions — Health Education; Myocardial Infarction; Emergencies

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- first aid and helping behaviour (Experimental): The helping behaviour training is given after 24 hours first aid training and aims to sensitise participants towards a helping reaction and teach participants how to deal with barriers to helping
  Interventions: Other: Helping behaviour curriculum
- first aid only (Active Comparator): This group receives training in first aid only without training in helping behaviour.
  Interventions: Other: First aid only curriculum

INTERVENTIONS:
Other: Helping behaviour curriculum — The objective of the helping behaviour curriculum is to sensitise participants to develop a helping reaction, and to teach participants how to deal with barriers to helping. The helping behaviour curriculum is being taught in 2hours.
  Arms: first aid and helping behaviour
Other: First aid only curriculum — Two hours training on first aid for alcohol and drug incidents
  Arms: first aid only

SUMMARY:
The objective of this study is to measure the effect of an innovative training programme on the help seeking behaviour and helping rates of bystanders in medical emergencies.

DETAILED DESCRIPTION:
A systematic review on the effects of first aid training concluded that training must also include ways to overcome obstacles to bystander intervention. This could lead to better help and higher helping rates in medical emergencies.

The objective of this paper is to measure the effect of an innovative training programme on the help seeking behaviour and helping rates of bystanders in medical emergencies. We chose to test the helping behaviour for acute myocardial infarction because it is an important cause of mortality and invalidity. While the victim is urgently in need of help, delay in seeking professional help is an important problem.

ELIGIBILITY:
Inclusion Criteria:

* Course participants that are 18 years or older

Exclusion Criteria:

* Course participants that are younger than 18 years
* Health care students
* Health care professionals

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2009-09; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Delay time for seeking help during deception experiment | within 4 weeks after the control or intervention training
  Time to seeking help was measured between the simulated patient grabbing the heart and the study participant opening the door to get help.

SECONDARY OUTCOMES:
Rate of helping during deception experiment | within 4 weeks after control or intervention training
  This refers to the number of participants that assessed the victim, or asked for help, or provided direct help to the victim during the test.
First aid self efficacy belief | within 15 minutes after experimental or control intervention
  scores on 6 questions related to helping behaviour barriers with the following structure: " I will do x (action) even if y (barrier)"
Impact of event | Within 15 minutes after deception experiment
  This indicates how shocking the study participants found the simulated emergency situation
State of mood | Within 15 minutes after deception experiment
  Indication of how study participants feel after being told about the deception.
Credibility of deception | Within 15 minutes after deception
  Indication of how credible study participants found the simulated emergency situation

CONTACTS AND LOCATIONS:
Overall Officials: Bert Aertgeerts, Principal Investigator — Academic Centre for General Practice, Catholic University Leuven
Locations (1):
- Belgian Red Cross-Flanders, Mechelen, Belgium

REFERENCES:
- [Background] Van de Velde S, Heselmans A, Roex A, Vandekerckhove P, Ramaekers D, Aertgeerts B. Effectiveness of nonresuscitative first aid training in laypersons: a systematic review. Ann Emerg Med. 2009 Sep;54(3):447-57, 457.e1-5. doi: 10.1016/j.annemergmed.2008.11.005. Epub 2009 Jan 21. PMID 19157654
- [Derived] Van de Velde S, Roex A, Vangronsveld K, Niezink L, Van Praet K, Heselmans A, Donceel P, Vandekerckhove P, Ramaekers D, Aertgeerts B. Can training improve laypersons helping behaviour in first aid? A randomised controlled deception trial. Emerg Med J. 2013 Apr;30(4):292-7. doi: 10.1136/emermed-2012-201128. Epub 2012 May 5. PMID 22562070